CLINICAL TRIAL: NCT00757549
Title: Comparison of FLT and FDG PET in the Evaluation of Response to Cetuximab, Cisplatin and Radiation Therapy in Advanced Head and Neck Malignancies or Response to Standard Chemo-radiotherapy in Esophageal Malignancies
Brief Title: 3'-Deoxy-3'-[18F] Fluorothymidine and Fludeoxyglucose F 18 PET Scans in Evaluating Response to Cetuximab, Cisplatin, and Radiation Therapy in Patients With Advanced Cancer of the Oropharynx, Larynx, or Hypopharynx
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Diagnostic
Other Study IDs: MC057M; P30CA015083 (NIH); MC057M (Other: Mayo Clinic Cancer Center); 08-002166 (Other: Mayo Clinic IRB); NCI-2009-01193 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-03

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Cisplatin; alovudine; Immunohistochemistry; Fluorodeoxyglucose F18; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: cetuximab
Drug: cisplatin
Genetic: TdT-mediated dUTP nick end labeling assay
Other: 3'-deoxy-3'-[18F]fluorothymidine
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Radiation: fludeoxyglucose F 18
Radiation: radiation therapy

SUMMARY:
RATIONALE: Diagnostic procedures, such as 3'-deoxy-3'-[18F] fluorothymidine (FLT) and fludeoxyglucose F 18 (FDG) PET scans, may help doctors predict a patient's response to treatment and help plan the best treatment.

PURPOSE: This pilot trial is studying FLT and FDG PET scans to see how well they evaluate response to cetuximab, cisplatin, and radiation therapy in patients with advanced cancer of the oropharynx, larynx, or hypopharynx.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess whether 3'-deoxy-3'-[18F] fluorothymidine (FLT) and fludeoxyglucose F 18 (FDG) PET scans can be used to identify patients with advanced squamous cell carcinoma of the oropharynx, larynx, or hypopharynx who have a biochemical response after 2 weeks of induction therapy with cetuximab.
* To assess whether FLT and FDG PET imaging-based response after 20-30 Gy of radiotherapy is predictive of disease control at 6 months after completion of therapy.

Secondary

* To assess whether FLT and FDG PET imaging-based response after cetuximab therapy and/or 20-30 Gy of radiotherapy is predictive of pathologic complete response in these patients.
* To assess whether FLT and FDG PET imaging-based response after cetuximab therapy and/or 20-30 Gy of radiotherapy is predictive of disease-free survival at 2 years in these patients.
* To correlate suppression of FLT uptake after cetuximab therapy with thymidine kinase 1 activity and/or expression, proliferation, microvessel density, apoptosis, and signaling pathway analyses.
* To correlate suppression of FDG uptake after cetuximab therapy with expression of hexokinases, glucose transporter proliferation, microvessel density, apoptosis, and signaling pathway analyses.
* To test and refine the ability of a novel commercial software package to quantify treatment-induced structural and functional/molecular volumetric and sub-volumetric change.
* To develop a working method for expressing change and predicting outcome.

OUTLINE: Patients receive cetuximab IV on days 1 and 8 of course 1. Beginning in course 2 and all subsequent courses, patients receive cetuximab IV and cisplatin IV over 2 hours on day 1 and undergo radiotherapy once daily 5 days a week for 7 weeks. Treatment repeats every 7 days for a total of 8 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo 3'-deoxy-3'-[18F] fluorothymidine and fludeoxyglucose F 18 (FDG) PET scans at baseline, after the second dose of cetuximab, after 20-30 Gy of radiotherapy, and then at 6 weeks and 6 months after completion of radiotherapy.

Patients undergo tumor tissue biopsies at baseline and after the first dose of cetuximab for correlative laboratory studies. Samples are analyzed for proliferation (Ki-67 labeling index), microvessel density (CD-31 staining), apoptosis (TUNEL assay and caspase-3 by IHC) signaling pathway (expression of EGFR, AKT, and MAPK by IHC), molecules affecting FDG uptake (expression of GLUT1, GLUT3, and hexokinase by IHC), and thymidine kinase 1 activity or expression.

After completion of study treatment, patients are followed every 3 months for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed squamous cell carcinoma of the oropharynx, larynx, or hypopharynx

  * Advanced disease
* Requires chemoradiotherapy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 16 weeks
* Weight loss ≤ 10% within the past 3 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 3 times ULN
* Hemoglobin ≥ 8 g/dL
* Creatinine clearance ≥ 40 mL/min
* No peripheral neuropathy ≥ grade 2
* No NYHA class III-IV heart disease
* No uncontrolled infection
* No poorly controlled diabetes that would limit the ability to obtain reliable fludeoxyglucose F 18 PET scan results
* No other severe underlying disease that, in the judgment of the investigator, would preclude study participation

PRIOR CONCURRENT THERAPY:

* More than 2 weeks since prior major surgery and recovered
* No prior radiotherapy to the planned treatment field
* No concurrent prophylactic filgrastim (G-CSF) or sargramostim (GM-CSF)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-09; Primary Completion 2011-08 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Percent change in the standard uptake value levels calculated for the identified volumes of interest for FLT and FDG PET scans from baseline to after 2 weeks of cetuximab therapy and from baseline to after 20-30 Gy of radiotherapy

SECONDARY OUTCOMES:
Quantified change values (after cetuximab therapy and after 20-30 Gy of radiotherapy) for the FLT and FDG PET scan-based topographic profiles created using the ImQuant software package

CONTACTS AND LOCATIONS:
Overall Officials: Jann N. Sarkaria, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States